CLINICAL TRIAL: NCT00202488
Title: The Effect of H. Pylori Infection on Iron Metabolism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry); Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-1807-B 03; RAB-EMR-420
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Iron Deficiency Anemia; Helicobacter Pylori Infection
Keywords: anemia, iron-deficiency; Helicobacter pylori
MeSH Terms: conditions — Anemia, Iron-Deficiency

INTERVENTIONS:
Drug: H. pylori treatment

SUMMARY:
The purpose of this study is to determine if Helicobacter pylori (H. pylori) gastritis results in abnormal iron metabolism in patients with iron deficiency anemia (IDA), and to determine if this is due to strain variations in the H. pylori organism.

DETAILED DESCRIPTION:
There is suggestive evidence that H. pylori gastritis (without peptic ulcer disease) is a cause of IDA. There have been individual case reports and case series describing patients with refractory IDA that resolved following successful H. pylori treatment. The effect of H. pylori on iron metabolism will be studied through specific aims: 1. To assess whether H. pylori results in abnormal oral iron absorption 2. To assess if differences in H. pylori strains are associated with iron deficiency due to: a. genetic differences in H. pylori strains or b. differences in the pattern of gastritis which could be due to host, bacterial or environmental factors 3. To assess if H. pylori infection results in storage of iron in the gastric mucosa and an elevated gastric iron concentration. The study will consist of three aspects: 1. Determining whether oral iron absorption is abnormal for H. pylori-positive IDA patients, and comparison of oral iron absorption for H. pylori positive and negative IDA patients. This will also include an experimental component in which oral iron absorption will be repeated after H. pylori treatment for H. pylori-infected IDA subjects (and after an equivalent time period for H. pylori negative controls to exclude changes in iron absorption that occur over time). 2. Comparison of H. pylori strain characteristics for IDA patients and non-anemic H. pylori-infected controls. Characterization of H. pylori strains will include: genetic analysis using a whole genome microarray technique that assesses the presence or absence of H. pylori genes, evaluation of expression of genes related to iron metabolism, and comparison of pattern of gastritis (pan gastritis vs. antrum-predominant). 3. Determination of whether H. pylori stores a significant quantity of iron in the gastric mucosa in vivo. This will be assessed by measuring the iron concentration in mucosal biopsy specimens and comparing results for H. pylori-infected IDA patients to H. pylori-uninfected IDA controls.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* iron deficiency anemia (IDA) defined as: Hgb < 14 g/L for men and 12 g/L for women, and a serum ferritin level less than 45 ug/L

Exclusion Criteria:

* Obvious non-GI cause of blood loss
* Chronic renal failure (BUN>60, Creatinine > 4)
* Hemolytic anemia, thalassemia, aplastic anemia
* Known alcoholism or cirrhosis of the liver
* Regular use (>3x weekly) of NSAIDS
* Prior gastric resection
* Celiac disease
* Known GI or hematologic malignancy
* Known inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39
Dates: Start 2002-11; Study Completion 2007-09

PRIMARY OUTCOMES:
Difference in iron absorption (Cmax) for H. pylori infected and uninfected IDA patients.
Change following H. pylori treatment in the iron absorption (Cmax) for H. pylori infected IDA patients.
Difference in the presence of genes related to iron metabolism for H. pylori-infected IDA patients vs. non-anemic controls.
Difference in gastritis pattern between H. pylori-infected IDA patients and non-anemic controls.

SECONDARY OUTCOMES:
Difference in gastritis severity between H. pylori-infected IDA patients and non-anemic controls.
Difference in gastric iron concentration.
Change in Hct and ferritin values following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: David Kearney, MD, Principal Investigator — University of Washington
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States